CLINICAL TRIAL: NCT02919033
Title: A Coordinated PCP-Cardiologist Telemedicine Model (PCTM) in China's Community Hypertension Care: Study Protocol for a Randomized Controlled Trial
Brief Title: Compare the Effects of Telemedicine Approach With Usual Care in Hypertension Management in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xu Lei (Other)
Responsible Party: Sponsor-Investigator, Xu Lei, Associate Chief, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SHDC12015308
Record Dates: First submitted 2016-09-23; First posted 2016-09-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Hypertension
Keywords: randomized controlled trial; telemedicine; hypertension; primary care; medication adherence
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual care (UC) (Placebo Comparator): Patients are managed by their PCPs at the registered CHCs as usual.
  Interventions: Other: Usual care
- Self-management (Experimental): * BP tele-monitor & App based self-management supports
  * Patient proficiency training
  Interventions: Device: Self-management
- PCTM intervention (Experimental): * BP tele-monitor & App-based self-management supports
  * Patient proficiency training
  * PCP & cardiologist training of using Web-based analytics
  * Proactive and interactive care by PCPs and cardiologists
  Interventions: Other: PCTM intervention

INTERVENTIONS:
Other: Usual care — The hypertension care of this arm complies with the national guideline and includes designated follow-ups by PCPs once every 1-3 months for stage-1 (≥ 140/90 mm Hg) hypertension patients, once every 1 month for stage-2 (≥ 160/100 mm Hg) and once every 2 weeks for stage-3 (≥ 180/110 mm Hg) patients.
  Arms: Usual care (UC)
Device: Self-management — * Usual care
  * Patients receive a BP telemedicine system developed by CareLinker Inc. (Shanghai, China) to facilitate BP self-management in addition to all the usual care components. The system consists of: 1) a BP tele-monitor with embedded GSM module that can upload BP readings; 2) a mobile App that allows patients to manually input healthcare data, display history BP measurements and lab test results, receive personalized lifestyle coaching contents and medication reminders, and communicate with PCPs through text-messaging.
  * All patients receive proficiency training in using the BP tele-monitor, and mobile App.
  Arms: Self-management
Other: PCTM intervention — * Usual care
  * Self-management
  * PCPs and cardiologists use the secure CareLinker website to review patient data including BP measurements, lab test results and medications in use and comorbidities. The auto analytics tools of the website reveal BP average, BP trend, and risk score of each patient. Text alerts of abnormal BP variability will be pushed to PCPs' App when they occur and proactive interventions including phone consultation and medication dosage adjustment will be offered. A case review session will be set once every 1-2 months for PCPs and cardiologists to exam patients' disease progresses. The proprietary web-based analytic module also produces automated individualized medication recommendations to PCPs.
  * PCPs and cardiologists receive training of the CareLinker website.
  Arms: PCTM intervention

SUMMARY:
This three arm study is to compare the effects of a coordinated PCP-Cardiologist Telemedicine Model (PCTM) with usual care and self-care in community hypertension management in China.

DETAILED DESCRIPTION:
Background: Hypertension is a major risk factor for cardiovascular diseases and its control rate has remained low worldwide. Studies have found that telemonitoring blood pressure (BP) helped control hypertension in randomized controlled trials. However, little is known about its effect in a structured primary care model in which primary care physicians (PCP) are partnering with cardiology specialists in electronic healthcare data sharing and medical interventions. This study aims to identify the effects of a coordinated PCP-Cardiologist model that applies telemedicine tools to facilitate community hypertension control in China.

Methods/Design: Hypertensive patients receiving care at four community healthcare centers (CHCs) that are academically affiliated to Shanghai Chest Hospital, Shanghai JiaoTong University are eligible if they have uncontrolled blood pressure in the previous three months and access to mobile internet. Study subjects are randomly assigned to three interventional groups: 1) usual care; 2) home-based BP tele-monitor with embedded GSM module and unlimited data plan, an App to access personal healthcare record and receive personalized lifestyle coaching contents, and proficiency training of their use; or 3) this plus coordinated PCP-Cardiologist care in which PCPs and cardiologists share data via a secure CareLinker website to determine interventional approaches. The primary outcome is mean change in systolic blood pressure (SBP) over a 12-month period. Secondary outcomes are changes of diastolic blood pressure (DBP), HbA1C, blood lipids, and medication adherence measured by the eight-item Morisky Medication Adherence Scale MMAS.

Discussion: This study will determine whether a coordinated PCP-Cardiologist Telemedicine Model (PCTM) that incorporates the lasted telemedicine technologies will improve hypertension care. Success of the model would help streamline the present community healthcare processes and impact a greater number of uncontrolled hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

1. age 21 years or older
2. a clinical diagnosis of hypertension with uncontrolled BP in the previous three months, currently taking or about to take anti-hypertensive medications
3. received high school or above level of education
4. active user of smart phone (Android or Apple) and mobile Apps
5. the average of three BP measurements during the screening visit at the CHC is ≥ 140/90 mm Hg, or ≥ 130/80 mm Hg if the patient has diabetes or renal diseases;
6. being able to give informed consent.

Exclusion Criteria:

* acute coronary syndrome
* heart failure
* cardiac arrhythmia
* stroke within the past three months
* renal failure
* cancer
* dementia, severe or acute psychiatric illness, pregnancy or intention to be pregnant in the next 18 months, and hospitalization within 3 months.
* additional exclusion criteria include participation in another clinical trial, arm
* circumference >32 centimeters that may affect the accuracy of BP measurement due to cuff size limit of the tele-monitor's, and unwillingness to comply with the 12 month intervention duration.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Changes in mean SBP | From baseline (T1) to 12 months (T3)
  The primary endpoint of the trial is changes in mean SBP from baseline (T1) to 12 months (T3) measured using the BP tele-monitor (Bliss BL928). The 12 months BP readings will be determined by taking the average of three BP measurements at the follow-up visit to the CHC. All BP data are collected and uploaded simultaneously to the trial database.

SECONDARY OUTCOMES:
Changes in mean DBP | From baseline (T1) to 12 months (T3)
  Changes of DBP will be determined at the same time as SBP, as described in the session of "Primary Outcome Measure"
Hypertension control rate | From baseline (T1) to 6 months (T2) and 12 months (T3)
  Hypertension control rate defined as BP < 140/90 mm Hg or < 130/80 mm Hg (patients of diabetes or renal diseases) following the national guidelines, and changes in measures related to hypertension complications (HbA1C, BMI, and lipid levels) from baseline (T1) to 6 months (T2) and 12 months (T3).
Anti-hypertensive medication adherence | At baseline (T1) and 12 months (T3).
  Adherence is assessed by self-report, eight-item Morisky Medication Adherence Scale MMAS modified to focus on BP drugs at baseline (T1) and 12 months (T3).

CONTACTS AND LOCATIONS:
Overall Officials: Lei Xu, Master, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hostpital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang G, Wang Y, Zeng Y, Gao GF, Liang X, Zhou M, Wan X, Yu S, Jiang Y, Naghavi M, Vos T, Wang H, Lopez AD, Murray CJ. Rapid health transition in China, 1990-2010: findings from the Global Burden of Disease Study 2010. Lancet. 2013 Jun 8;381(9882):1987-2015. doi: 10.1016/S0140-6736(13)61097-1. PMID 23746901
- [Background] Law MR, Morris JK, Wald NJ. Use of blood pressure lowering drugs in the prevention of cardiovascular disease: meta-analysis of 147 randomised trials in the context of expectations from prospective epidemiological studies. BMJ. 2009 May 19;338:b1665. doi: 10.1136/bmj.b1665. PMID 19454737
- [Background] Dickinson HO, Mason JM, Nicolson DJ, Campbell F, Beyer FR, Cook JV, Williams B, Ford GA. Lifestyle interventions to reduce raised blood pressure: a systematic review of randomized controlled trials. J Hypertens. 2006 Feb;24(2):215-33. doi: 10.1097/01.hjh.0000199800.72563.26. PMID 16508562
- [Background] Blood Pressure Lowering Treatment Trialists' Collaboration. Blood pressure-lowering treatment based on cardiovascular risk: a meta-analysis of individual patient data. Lancet. 2014 Aug 16;384(9943):591-598. doi: 10.1016/S0140-6736(14)61212-5. PMID 25131978
- [Background] Kumar N, Khunger M, Gupta A, Garg N. A content analysis of smartphone-based applications for hypertension management. J Am Soc Hypertens. 2015 Feb;9(2):130-6. doi: 10.1016/j.jash.2014.12.001. Epub 2014 Dec 11. PMID 25660364
- [Background] Quinn CC, Clough SS, Minor JM, Lender D, Okafor MC, Gruber-Baldini A. WellDoc mobile diabetes management randomized controlled trial: change in clinical and behavioral outcomes and patient and physician satisfaction. Diabetes Technol Ther. 2008 Jun;10(3):160-8. doi: 10.1089/dia.2008.0283. PMID 18473689
- [Background] Pfaeffli Dale L, Whittaker R, Jiang Y, Stewart R, Rolleston A, Maddison R. Text Message and Internet Support for Coronary Heart Disease Self-Management: Results From the Text4Heart Randomized Controlled Trial. J Med Internet Res. 2015 Oct 21;17(10):e237. doi: 10.2196/jmir.4944. PMID 26490012
- [Background] Fernandez-Granero MA, Sanchez-Morillo D, Leon-Jimenez A. Computerised Analysis of Telemonitored Respiratory Sounds for Predicting Acute Exacerbations of COPD. Sensors (Basel). 2015 Oct 23;15(10):26978-96. doi: 10.3390/s151026978. PMID 26512667
- [Background] Quinn CC, Shardell MD, Terrin ML, Barr EA, Ballew SH, Gruber-Baldini AL. Cluster-randomized trial of a mobile phone personalized behavioral intervention for blood glucose control. Diabetes Care. 2011 Sep;34(9):1934-42. doi: 10.2337/dc11-0366. Epub 2011 Jul 25. PMID 21788632
- [Background] Omboni S, Caserini M, Coronetti C. Telemedicine and M-Health in Hypertension Management: Technologies, Applications and Clinical Evidence. High Blood Press Cardiovasc Prev. 2016 Sep;23(3):187-96. doi: 10.1007/s40292-016-0143-6. Epub 2016 Apr 12. PMID 27072129
- [Background] Omboni S, Gazzola T, Carabelli G, Parati G. Clinical usefulness and cost effectiveness of home blood pressure telemonitoring: meta-analysis of randomized controlled studies. J Hypertens. 2013 Mar;31(3):455-67; discussion 467-8. doi: 10.1097/HJH.0b013e32835ca8dd. PMID 23299557
- [Background] Quinn CC, Gruber-Baldini AL, Shardell M, Weed K, Clough SS, Peeples M, Terrin M, Bronich-Hall L, Barr E, Lender D. Mobile diabetes intervention study: testing a personalized treatment/behavioral communication intervention for blood glucose control. Contemp Clin Trials. 2009 Jul;30(4):334-46. doi: 10.1016/j.cct.2009.02.004. Epub 2009 Feb 27. PMID 19250979
- [Background] Quinn CC, Sareh PL, Shardell ML, Terrin ML, Barr EA, Gruber-Baldini AL. Mobile Diabetes Intervention for Glycemic Control: Impact on Physician Prescribing. J Diabetes Sci Technol. 2014 Mar;8(2):362-370. doi: 10.1177/1932296813514503. Epub 2014 Feb 5. PMID 24876589
- [Background] Quinn CC, Shardell MD, Terrin ML, Barr EA, Park D, Shaikh F, Guralnik JM, Gruber-Baldini AL. Mobile Diabetes Intervention for Glycemic Control in 45- to 64-Year-Old Persons With Type 2 Diabetes. J Appl Gerontol. 2016 Feb;35(2):227-43. doi: 10.1177/0733464814542611. Epub 2014 Aug 6. PMID 25098253
- [Background] Margolis KL, Asche SE, Bergdall AR, Dehmer SP, Maciosek MV, Nyboer RA, O'Connor PJ, Pawloski PA, Sperl-Hillen JM, Trower NK, Tucker AD, Green BB. A Successful Multifaceted Trial to Improve Hypertension Control in Primary Care: Why Did it Work? J Gen Intern Med. 2015 Nov;30(11):1665-72. doi: 10.1007/s11606-015-3355-x. PMID 25952653
- [Background] O'Connor PJ, Schmittdiel JA, Pathak RD, Harris RI, Newton KM, Ohnsorg KA, Heisler M, Sterrett AT, Xu S, Dyer WT, Raebel MA, Thomas A, Schroeder EB, Desai JR, Steiner JF. Randomized trial of telephone outreach to improve medication adherence and metabolic control in adults with diabetes. Diabetes Care. 2014 Dec;37(12):3317-24. doi: 10.2337/dc14-0596. Epub 2014 Oct 14. PMID 25315207
- [Background] Xu L, Zhang Y, Chen Y, Li YJ, Chen D, Wang T, Zhang HG, Qu WH, Liu K: The role of pharmacist-led hypertension management in China's community medical care service: a retrospective analysis of real-world big-data samples. Precision Medicine in Cardiology 2016, 1(1):19-26.
- [Background] Oliveira-Filho AD, Barreto-Filho JA, Neves SJ, Lyra Junior DP. Association between the 8-item Morisky Medication Adherence Scale (MMAS-8) and blood pressure control. Arq Bras Cardiol. 2012 Jul;99(1):649-58. doi: 10.1590/s0066-782x2012005000053. Epub 2012 Jun 7. English, Portuguese. PMID 22688844
- [Background] Liu LS; Writing Group of 2010 Chinese Guidelines for the Management of Hypertension. [2010 Chinese guidelines for the management of hypertension]. Zhonghua Xin Xue Guan Bing Za Zhi. 2011 Jul;39(7):579-615. Chinese. PMID 22088239
- [Background] Zhang HG, Liu K, Kong WJ, Tian F, Yang YR, Feng C, Wang T, Chen Q: A mobile health solution for chronic disease managment at retail pharmacy. IEEE Healthcom'16 2016, Sep(14).
- [Background] Wu Y, Liu X, Li X, Li Y, Zhao L, Chen Z, Li Y, Rao X, Zhou B, Detrano R, Liu K; USA-PRC Collaborative Study of Cardiovascular and Cardiopulmonary Epidemiology Research Group; China Multicenter Collaborative Study of Cardiovascular Epidemiology Research Group. Estimation of 10-year risk of fatal and nonfatal ischemic cardiovascular diseases in Chinese adults. Circulation. 2006 Nov 21;114(21):2217-25. doi: 10.1161/CIRCULATIONAHA.105.607499. Epub 2006 Nov 6. PMID 17088464
- [Background] Collaborative G: A study on evaluation of the risk of ischemic cardiovascular diseases in Chinese and the development of simplified tools for the evaluation. Chinese Journal of Cardiology 2003, 12.
- [Background] Li LM, Rao KQ, Kong LZ, Yao CH, Xiang HD, Zhai FY, Ma GS, Yang XG; Technical Working Group of China National Nutrition and Health Survey. [A description on the Chinese national nutrition and health survey in 2002]. Zhonghua Liu Xing Bing Xue Za Zhi. 2005 Jul;26(7):478-84. Chinese. PMID 16334996
- [Background] Sheng CS, Liu M, Kang YY, Wei FF, Zhang L, Li GL, Dong Q, Huang QF, Li Y, Wang JG. Prevalence, awareness, treatment and control of hypertension in elderly Chinese. Hypertens Res. 2013 Sep;36(9):824-8. doi: 10.1038/hr.2013.57. Epub 2013 Jun 13. PMID 23759756
- [Background] Wang L, Kong L, Wu F, Bai Y, Burton R. Preventing chronic diseases in China. Lancet. 2005 Nov 19;366(9499):1821-4. doi: 10.1016/S0140-6736(05)67344-8. PMID 16298221
- [Background] Yang G, Kong L, Zhao W, Wan X, Zhai Y, Chen LC, Koplan JP. Emergence of chronic non-communicable diseases in China. Lancet. 2008 Nov 8;372(9650):1697-705. doi: 10.1016/S0140-6736(08)61366-5. Epub 2008 Oct 17. PMID 18930526
- [Background] Hallberg I, Taft C, Ranerup A, Bengtsson U, Hoffmann M, Hofer S, Kasperowski D, Makitalo A, Lundin M, Ring L, Rosenqvist U, Kjellgren K. Phases in development of an interactive mobile phone-based system to support self-management of hypertension. Integr Blood Press Control. 2014 May 7;7:19-28. doi: 10.2147/IBPC.S59030. eCollection 2014. PMID 24910510
- [Background] Zullig LL, Melnyk SD, Goldstein K, Shaw RJ, Bosworth HB. The role of home blood pressure telemonitoring in managing hypertensive populations. Curr Hypertens Rep. 2013 Aug;15(4):346-55. doi: 10.1007/s11906-013-0351-6. PMID 23625207
- [Background] Kirwan M, Vandelanotte C, Fenning A, Duncan MJ. Diabetes self-management smartphone application for adults with type 1 diabetes: randomized controlled trial. J Med Internet Res. 2013 Nov 13;15(11):e235. doi: 10.2196/jmir.2588. PMID 24225149
- [Background] Logan AG, Irvine MJ, McIsaac WJ, Tisler A, Rossos PG, Easty A, Feig DS, Cafazzo JA. Effect of home blood pressure telemonitoring with self-care support on uncontrolled systolic hypertension in diabetics. Hypertension. 2012 Jul;60(1):51-7. doi: 10.1161/HYPERTENSIONAHA.111.188409. Epub 2012 May 21. PMID 22615116
- [Background] Stoddart A, Hanley J, Wild S, Pagliari C, Paterson M, Lewis S, Sheikh A, Krishan A, Padfield P, McKinstry B. Telemonitoring-based service redesign for the management of uncontrolled hypertension (HITS): cost and cost-effectiveness analysis of a randomised controlled trial. BMJ Open. 2013 May 28;3(5):e002681. doi: 10.1136/bmjopen-2013-002681. PMID 23793650
- [Background] Thiboutot J, Sciamanna CN, Falkner B, Kephart DK, Stuckey HL, Adelman AM, Curry WJ, Lehman EB. Effects of a web-based patient activation intervention to overcome clinical inertia on blood pressure control: cluster randomized controlled trial. J Med Internet Res. 2013 Sep 4;15(9):e158. doi: 10.2196/jmir.2298. PMID 24004475
- [Background] Kim JY, Wineinger NE, Steinhubl SR. The Influence of Wireless Self-Monitoring Program on the Relationship Between Patient Activation and Health Behaviors, Medication Adherence, and Blood Pressure Levels in Hypertensive Patients: A Substudy of a Randomized Controlled Trial. J Med Internet Res. 2016 Jun 22;18(6):e116. doi: 10.2196/jmir.5429. PMID 27334418
- [Background] Hosseininasab M, Jahangard-Rafsanjani Z, Mohagheghi A, Sarayani A, Rashidian A, Javadi M, Ahmadvand A, Hadjibabaie M, Gholami K. Self-monitoring of blood pressure for improving adherence to antihypertensive medicines and blood pressure control: a randomized controlled trial. Am J Hypertens. 2014 Nov;27(11):1339-45. doi: 10.1093/ajh/hpu062. Epub 2014 Apr 26. PMID 24771706
- [Background] McManus RJ, Mant J, Bray EP, Holder R, Jones MI, Greenfield S, Kaambwa B, Banting M, Bryan S, Little P, Williams B, Hobbs FD. Telemonitoring and self-management in the control of hypertension (TASMINH2): a randomised controlled trial. Lancet. 2010 Jul 17;376(9736):163-72. doi: 10.1016/S0140-6736(10)60964-6. Epub 2010 Jul 8. PMID 20619448
- [Background] Hirsch JD, Steers N, Adler DS, Kuo GM, Morello CM, Lang M, Singh RF, Wood Y, Kaplan RM, Mangione CM. Primary care-based, pharmacist-physician collaborative medication-therapy management of hypertension: a randomized, pragmatic trial. Clin Ther. 2014 Sep 1;36(9):1244-54. doi: 10.1016/j.clinthera.2014.06.030. Epub 2014 Jul 30. PMID 25085406
- [Background] Carter BL, Ardery G, Dawson JD, James PA, Bergus GR, Doucette WR, Chrischilles EA, Franciscus CL, Xu Y. Physician and pharmacist collaboration to improve blood pressure control. Arch Intern Med. 2009 Nov 23;169(21):1996-2002. doi: 10.1001/archinternmed.2009.358. PMID 19933962
- [Background] Carter BL, Coffey CS, Ardery G, Uribe L, Ecklund D, James P, Egan B, Vander Weg M, Chrischilles E, Vaughn T. Cluster-randomized trial of a physician/pharmacist collaborative model to improve blood pressure control. Circ Cardiovasc Qual Outcomes. 2015 May;8(3):235-43. doi: 10.1161/CIRCOUTCOMES.114.001283. Epub 2015 Mar 24. PMID 25805647
- [Background] O'Neill JL, Cunningham TL, Wiitala WL, Bartley EP. Collaborative hypertension case management by registered nurses and clinical pharmacy specialists within the Patient Aligned Care Teams (PACT) model. J Gen Intern Med. 2014 Jul;29 Suppl 2(Suppl 2):S675-81. doi: 10.1007/s11606-014-2774-4. PMID 24715403
- [Background] Hunt JS, Siemienczuk J, Pape G, Rozenfeld Y, MacKay J, LeBlanc BH, Touchette D. A randomized controlled trial of team-based care: impact of physician-pharmacist collaboration on uncontrolled hypertension. J Gen Intern Med. 2008 Dec;23(12):1966-72. doi: 10.1007/s11606-008-0791-x. Epub 2008 Sep 25. PMID 18815843
- [Background] Qudah B, Albsoul-Younes A, Alawa E, Mehyar N. Role of clinical pharmacist in the management of blood pressure in dialysis patients. Int J Clin Pharm. 2016 Aug;38(4):931-40. doi: 10.1007/s11096-016-0317-2. Epub 2016 May 18. PMID 27194097
- [Background] Green BB, Cook AJ, Ralston JD, Fishman PA, Catz SL, Carlson J, Carrell D, Tyll L, Larson EB, Thompson RS. Effectiveness of home blood pressure monitoring, Web communication, and pharmacist care on hypertension control: a randomized controlled trial. JAMA. 2008 Jun 25;299(24):2857-67. doi: 10.1001/jama.299.24.2857. PMID 18577730
- [Background] Magid DJ, Olson KL, Billups SJ, Wagner NM, Lyons EE, Kroner BA. A pharmacist-led, American Heart Association Heart360 Web-enabled home blood pressure monitoring program. Circ Cardiovasc Qual Outcomes. 2013 Mar 1;6(2):157-63. doi: 10.1161/CIRCOUTCOMES.112.968172. Epub 2013 Mar 5. PMID 23463811
- [Background] Green BB, Anderson ML, Ralston JD, Catz SL, Cook AJ. Blood pressure 1 year after completion of web-based pharmacist care. JAMA Intern Med. 2013 Jul 8;173(13):1250-2. doi: 10.1001/jamainternmed.2013.1037. No abstract available. PMID 23689927
- [Background] Margolis KL, Asche SE, Bergdall AR, Dehmer SP, Groen SE, Kadrmas HM, Kerby TJ, Klotzle KJ, Maciosek MV, Michels RD, O'Connor PJ, Pritchard RA, Sekenski JL, Sperl-Hillen JM, Trower NK. Effect of home blood pressure telemonitoring and pharmacist management on blood pressure control: a cluster randomized clinical trial. JAMA. 2013 Jul 3;310(1):46-56. doi: 10.1001/jama.2013.6549. PMID 23821088
- [Background] Omboni S, Sala E. The pharmacist and the management of arterial hypertension: the role of blood pressure monitoring and telemonitoring. Expert Rev Cardiovasc Ther. 2015 Feb;13(2):209-21. doi: 10.1586/14779072.2015.1001368. Epub 2015 Jan 12. PMID 25578090
- [Background] Lee P, Liu JC, Hsieh MH, Hao WR, Tseng YT, Liu SH, Lin YK, Sung LC, Huang JH, Yang HY, Ye JS, Zheng HS, Hsu MH, Syed-Abdul S, Lu R, Nguyen PA, Iqbal U, Huang CW, Jian WS, Li YC. Cloud-based BP system integrated with CPOE improves self-management of the hypertensive patients: A randomized controlled trial. Comput Methods Programs Biomed. 2016 Aug;132:105-13. doi: 10.1016/j.cmpb.2016.04.003. Epub 2016 Apr 7. PMID 27282232
- [Background] Omboni S, Guarda A. Impact of home blood pressure telemonitoring and blood pressure control: a meta-analysis of randomized controlled studies. Am J Hypertens. 2011 Sep;24(9):989-98. doi: 10.1038/ajh.2011.100. Epub 2011 Jun 9. PMID 21654858
- [Background] van Vugt M, de Wit M, Cleijne WH, Snoek FJ. Use of behavioral change techniques in web-based self-management programs for type 2 diabetes patients: systematic review. J Med Internet Res. 2013 Dec 13;15(12):e279. doi: 10.2196/jmir.2800. PMID 24334230
- [Background] AbuDagga A, Resnick HE, Alwan M. Impact of blood pressure telemonitoring on hypertension outcomes: a literature review. Telemed J E Health. 2010 Sep;16(7):830-8. doi: 10.1089/tmj.2010.0015. PMID 20815751
- [Background] Santschi V, Chiolero A, Colosimo AL, Platt RW, Taffe P, Burnier M, Burnand B, Paradis G. Improving blood pressure control through pharmacist interventions: a meta-analysis of randomized controlled trials. J Am Heart Assoc. 2014 Apr 10;3(2):e000718. doi: 10.1161/JAHA.113.000718. PMID 24721801
- [Derived] Xu L, Fang WY, Zhu F, Zhang HG, Liu K. A coordinated PCP-Cardiologist Telemedicine Model (PCTM) in China's community hypertension care: study protocol for a randomized controlled trial. Trials. 2017 May 25;18(1):236. doi: 10.1186/s13063-017-1970-z. PMID 28545514